CLINICAL TRIAL: NCT06976307
Title: Development of an Adaptive Treatment Strategy for Weight Loss in People With Prediabetes Using a Sequential Multiple Assignment Randomized Trial
Brief Title: Development of an Inclusive Adaptive Treatment Strategy for Weight Loss in People With Prediabetes Using a Sequential Multiple Assignment Randomized Trial
Acronym: iADAPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Christine Ferguson, PhD, RD, LD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300006816-sub-study; CEDHARS (Other Grant/Funding Number: Center for Engagement in Disability Health and Rehabilitation Sciences (CEDHARS); University of Alabama at Birmingham)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Disabilities; Obesity and Overweight; Prediabetes
Keywords: SMART; diet; exercise; weight loss; disabilities
MeSH Terms: conditions — Obesity; Overweight; Prediabetic State; Motor Activity; Weight Loss | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Carbohydrate Diet (Experimental): Enrollment in a group-based behavioral weight loss intervention based on the Diabetes Prevention Program curriculum with high carbohydrate diet plan.
  Interventions: Behavioral: High Carbohydrate Diet
- Reduced Carbohydrate Diet (Experimental): Enrollment in a group-based behavioral weight loss intervention based on the Diabetes Prevention Program curriculum with reduced carbohydrate diet plan.
  Interventions: Behavioral: Reduced Carbohydrate Diet

INTERVENTIONS:
Behavioral: High Carbohydrate Diet — Participants randomized to this group will participate in a group-based weight behavioral management program and consume a high carbohydrate (HC) diet. Because this protocol uses a sequential, multiple assignment, randomized trial (SMART) design, response will be assessed at week 4. Responders will continue with their 1st stage assignment for the remainder of the study. Non-responders will be randomized to 2nd stage intervention of either combine HC diet with time-restricted eating (TRE) or HC diet with additional exercise counseling and support.
  Arms: High Carbohydrate Diet
Behavioral: Reduced Carbohydrate Diet — Participants randomized to this group will participate in a group-based behavioral weight management program and consume a reduced carbohydrate (RC) diet. Because this is a sequential, multiple assignment, randomized trial (SMART) design, response will be assessed at week 4. Responders will continue with their 1st stage assignment for the remainder of the study. Non-responders will be randomized to 2nd stage intervention of either combine RC diet with time-restricted eating (TRE) or RC diet with additional exercise counseling and support.
  Arms: Reduced Carbohydrate Diet

SUMMARY:
This is a sub-study to NCT04745572 to include a new cohort of participants with disabilities. This 16-week study will use an experimental approach called the Sequential Multiple Assignment Randomized Trial to help determine which combination and sequence of weight loss program features are most effective in people who are at risk for type 2 diabetes. Participants in the study will be initially randomized to consume either a high or reduced carbohydrate diet. After 4 weeks, participants will be identified as Responders (greater than or equal to 2.5% weight loss) or Non-Responders (less than 2.5% weight loss). Responders will continue with their initial randomized group for the remainder of the trial. Non-responders will be re-randomized to 2nd stage interventions of either including additional exercise counseling and training or beginning a time restricted eating protocol for the remainder of the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* BMI of 27 kg/m2 or greater for ambulatory individuals and 22 kg/m2 for individuals with spinal cord injury. Adjustments will be calculated for those with amputations and/or limb indifference
* at risk for developing type 2 diabetes (prediabetes)
* One or more physical or mobility disabilities
* Stable medication type and dosage for 3 or more months for medications likely to affect body weight and/or appetite
* Willing to complete requirements for participation

Exclusion Criteria:

* Pregnant, planning to become pregnant or breastfeeding
* Currently taking medication(s) for weight loss
* Medical history of Type 1 or 2 Diabetes, using exogenous insulin, using prescription or OTC weight loss medications within the past 3 months, current alcohol or drug abuse or dependence, smoker with unstable habits in the past 3 months, pacemaker or other life-threatening medical implant, eating disorder(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in glucose | Baseline & Week 16
  Serum glucose will be measured in a fasted state.
Changes in body weight | Baseline, Week4, and Week 16
  Measured on validated digital scale

SECONDARY OUTCOMES:
Changes in fat mass | Baseline & Week 16
  As measured by dual-energy X-ray absorptiometry (DEXA)
Change in insulin | Baseline & Week 16
  Serum insulin will be measured in a fasted state.
Changes in lipids | Baseline & Week 16
  Fasting serum concentrations of total cholesterol, HDL cholesterol, triglycerides, and LDL cholesterol
Changes in QUICKI index | Baseline & Week 16
  Predictor of insulin resistance that will be calculated from glucose and insulin measures
Changes in overall strength | Baseline & Week 16
  As measured by hand grip dynamometry
Changes in aerobic fitness | Baseline & Week 16
  As measured by graded exercise test using arm crank

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ferguson, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Wellness Health and Research Facility (WHARF), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No